CLINICAL TRIAL: NCT05572060
Title: Effect of Metformin Use on Mortality in Diabetic and Non Diabetic Patients With Sepsis and Septic Shock.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Khaled Ahmed Abodeef, anesthesiology and ICU resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Metformin use in sepsis
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C: (n=25) control. (Active Comparator): patients will receive standardized protocol without receiving metformin.
  Interventions: Other: standardized protocol
- Group D: (n=25) diabetic patients. (Active Comparator): diabetic patients will receive standardized protocol and receiving metformin 500 mg every 8 hours since admission regardless of their random blood sugar with measurement of random blood sugar every hour and dextrose 25% infusion will be used if needed and also insulin infusion will be used when appropriate with target random blood sugar 140-180 in diabetic patients.
  Interventions: Drug: Metformin; Other: standardized protocol
- Group ND: (n=25) non-diabetic patients. (Active Comparator): patients will receive standardized protocol and receiving metformin 500 mg every 8 hours since admission regardless of their random blood sugar with measurement of random blood sugar every hour and dextrose 25% infusion will be used if needed and also insulin infusion will be used when appropriate with target random blood sugar 100-140 in non diabetic patients.
  Interventions: Drug: Metformin; Other: standardized protocol

INTERVENTIONS:
Drug: Metformin — Patient screening will be done using SOFA scoring and NEWS Supplemental oxygen will be supplied. Intubation and mechanical ventilation may be required Venous access will be established.CBC, chemistries, liver function tests,coagulation studies ,Peripheral blood cultures, urinalysis, microbiological cultures from suspected sources (eg, sputum, urine,etc),(ABG) and serum lactate will be obtained Crystalloids will be given at 30 mL/kg, started by one hour and completed within three hours Empiric antibiotic therapy is targeted at the suspected organism(s) In patients with lactic acidosis and severe acidemia, Sodium bicarbonate will be used to maintain the arterial pH above 7.15 In patients having persistent hypoperfusion vasopressors will be added Evaluation of volume status will be done using straight leg raising test and ultrasound guided IVC collapsibility index Plasma rennin, serum lactate and IL6 concentrations will be measured on admission and at one week.
  Arms: Group D: (n=25) diabetic patients.; Group ND: (n=25) non-diabetic patients.
Other: standardized protocol — standardized protocol

SUMMARY:
We aimed to determine if metformin use in both diabetic and non diabetic patients with sepsis and septic shock affects 28 day mortality and its effect on inflammatory markers. Plasma rennin, serum lactate concentration and IL6 will be measured for predicting 28 days in-hospital mortality in patients with sepsis.

DETAILED DESCRIPTION:
Sepsis, is a life-threatening condition arises when the body's response to infection causes injury to its own tissues, followed by suppression of the immune system. Signs and symptoms include fever, increased heart rate, increased breathing rate, and confusion.There may be symptoms of a specific infection, such as cough, or painful urination.

Sepsis is caused by many organisms including bacteria, viruses and fungi. . Risk factors include extreme of ages, a weakened immune system. Previously, a sepsis diagnosis required the presence of at least two systemic inflammatory response syndrome criteria.

Sepsis requires immediate treatment with intravenous fluids and antimicrobials in ICU. If fluids is not enough to maintain blood pressure, the use of medications that raise blood pressure becomes necessary. Mechanical ventilation and dialysis may be needed. A central venous catheter and an arterial catheter may be placed. corticosteroid use is controversial.

Metformin is a biguanide antihyperglycemic agent. It works by decreasing glucose production in the liver, by increasing the insulin sensitivity of body tissues, and by increasing GDF15 secretion, which reduces appetite.

Metformin is a first-line therapy for type 2 diabetes mellitus, taken by mouth and well tolerated. Common adverse effects include diarrhea, nausea, and abdominal pain.

Metformin inhibit pathways linked to inflammation, immune reactions, mammalian target of rapamycin (mTOR) signaling, and cell senescence. Some of the changes were confirmed by Western blot. Therefore, metformin prevented part of the deleterious actions of pro-inflammatory cytokines in human β-cells, which was accompanied by islet proteome modifications.

ELIGIBILITY:
Inclusion Criteria:

* both sexes aged ≥18 years old complaining of sepsis or septic shock with anticipated stay >24 hours, and signed informed consent by patient or next-of-kin.

Exclusion Criteria:

* Age less than 18 years old, chronic kidney disease stage IV/V (baseline eGFR <30ml/min/1.73m2), patients with acute coronary syndrome, or do not resuscitate order. Patients could be enrolled at any point during their admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
28 day Mortality. | 28 day.
  death within 28 day of sepsis and septic shock where the occurrence of sepsis is hour 0 day 0.

SECONDARY OUTCOMES:
Plasma rennin concentration (pg/ml) will be measured on admission and at one week. | On admission and at 1 week after admission.
IL6 concentration (ng/ml) will be measured on admission and at one week. | On admission and at 1 week after admission.
  Level of inflammatory mediators on admission and at 1 week after admission.
Serum lactate concentration (mmol/L) will be measured on admission and at one week. | On admission and at 1 week after admission.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Khaled Ahmed Abodeef, resident, Study Chair — Assiut University; Abualauon Mohamed Abedalmohsen, MD, Study Director — Assiut University; Nagwa Mostafa Ibrahim, MD, Principal Investigator — Assiut University

REFERENCES:
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Deutschman CS, Tracey KJ. Sepsis: current dogma and new perspectives. Immunity. 2014 Apr 17;40(4):463-75. doi: 10.1016/j.immuni.2014.04.001. PMID 24745331
- [Background] Sehgal M, Ladd HJ, Totapally B. Trends in Epidemiology and Microbiology of Severe Sepsis and Septic Shock in Children. Hosp Pediatr. 2020 Dec;10(12):1021-1030. doi: 10.1542/hpeds.2020-0174. PMID 33208389
- [Background] Annane D, Bellissant E, Bollaert PE, Briegel J, Keh D, Kupfer Y, Pirracchio R, Rochwerg B. Corticosteroids for treating sepsis in children and adults. Cochrane Database Syst Rev. 2019 Dec 6;12(12):CD002243. doi: 10.1002/14651858.CD002243.pub4. PMID 31808551
- [Background] Giusti L, Tesi M, Ciregia F, Marselli L, Zallocco L, Suleiman M, De Luca C, Del Guerra S, Zuccarini M, Trerotola M, Eizirik DL, Cnop M, Mazzoni MR, Marchetti P, Lucacchini A, Ronci M. The Protective Action of Metformin against Pro-Inflammatory Cytokine-Induced Human Islet Cell Damage and the Mechanisms Involved. Cells. 2022 Aug 8;11(15):2465. doi: 10.3390/cells11152465. PMID 35954309
- [Background] Raith EP, Udy AA, Bailey M, McGloughlin S, MacIsaac C, Bellomo R, Pilcher DV; Australian and New Zealand Intensive Care Society (ANZICS) Centre for Outcomes and Resource Evaluation (CORE). Prognostic Accuracy of the SOFA Score, SIRS Criteria, and qSOFA Score for In-Hospital Mortality Among Adults With Suspected Infection Admitted to the Intensive Care Unit. JAMA. 2017 Jan 17;317(3):290-300. doi: 10.1001/jama.2016.20328. PMID 28114553